CLINICAL TRIAL: NCT01311193
Title: Circadian Sleep-wake Cycles, Well-being and Light Therapy in Borderline Personality Disorder
Brief Title: Circadian Sleep-wake Cycles and Light Therapy in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Velux Fonden (Other); Lumie UK (Unknown)
Other Study IDs: Velux-425
Record Dates: First submitted 2011-03-03; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Borderline Personality Disorder; Sleep Disturbances; Depression
Keywords: Circadian rhythms; Sleep-wake cycles; Melatonin; Borderline Personality Disorder; Light therapy
MeSH Terms: conditions — Borderline Personality Disorder; Parasomnias; Depression | interventions — Phototherapy

ARMS (1):
- light therapy (Experimental): Morning bright light treatment (at 8000 lux for 40min, daily during 3 weeks)
  Interventions: Other: light therapy

INTERVENTIONS:
Other: light therapy — early morning exposures to bright light, 8000lux for 40min, daily during 3 weeks

SUMMARY:
Individuals with borderline personality disorder (BPD) frequently suffer from emotional instability, daytime fatigue and sleep disturbances. The investigators examined circadian rhythms, sleep and well-being in women with BPD under their habitual life conditions with and without light treatment.

Treated women diagnosed with BPD were investigated during 3 weeks without and 3 weeks with morning LT. Rest-activity cycles were continuously measured using wrist actigraphy, together with proximal skin temperature. Saliva samples were collected weekly to determine the diurnal melatonin rhythm. A range of self-ratings and questionnaires were used to assess depression and clinical state throughout the 6-week protocol. Ten matched healthy women followed the same 6-week protocol without light treatment.

ELIGIBILITY:
Inclusion Criteria:

* Borderline Personality Disorder (DSM IV-criteria)
* German-speaking
* normal ocular function

Exclusion Criteria:

* lack of compliance

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Christian Cajochen, PhD, Principal Investigator — Centre for Chronobiology, Psychiatric Hospital, University of Basel
Locations (1):
- Centre for Chronobiology, Psychiatric Hospital, University of Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- See also: Related Info — http://www.chronobiology.ch